CLINICAL TRIAL: NCT01539174
Title: A Phase II Study of Rituximab Intense Dosing With CHOP-21 (RID-CHOP) in Patients With Previously Untreated High or High-Intermediate Risk IPI (3-5) Diffuse Large B-Cell Lymphoma (DLBCL)
Brief Title: Rituximab and Combination Chemotherapy in Treating Patients With Previously Untreated High- or High-Intermediate-Risk Diffuse Large B-Cell Lymphoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No Funding Source and Competing Trials
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OER-HM-039; NCI-2011-03309 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-02-15; First posted 2012-02-27 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Contiguous Stage II Adult Diffuse Large Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Large Cell Lymphoma; Stage I Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (monoclonal antibody, combination chemotherapy) (Experimental): Patients receive rituximab IV on days 0, 1, 4, 8, and 15 of course 1; days 1, 8, and 15 of course 2; and day 1 of all subsequent courses. Patients also receive CHOP chemotherapy comprising cyclophosphamide IV, doxorubicin hydrochloride IV, and vincristine sulfate IV on day 1, and prednisone PO on days 1-5. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: rituximab; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: vincristine sulfate; Drug: prednisone; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: doxorubicin hydrochloride — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Drug: vincristine sulfate — Given IV
  Other Names: leurocristine sulfate; VCR; Vincasar PFS
Drug: prednisone — Given PO
  Other Names: DeCortin; Deltra
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase II trial studies how well giving rituximab together with combination chemotherapy works in treating patients with previously untreated high- or high-intermediate-risk diffuse large B-cell lymphoma (DLBCL). Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy, such as cyclophosphamide, doxorubicin hydrochloride, vincristine sulfate, and prednisone (CHOP), work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug, combination chemotherapy, may kill more cancer cells. Giving rituximab together with combination chemotherapy together may be an effective treatment for DLBCL

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate 1 year progression-free survival (PFS) following treatment with rituximab intense dosing and CHOP-21 (RID-CHOP) in previously untreated patients with high risk (International Prognostic Index [IPI] 3-5) DLBCL.

SECONDARY OBJECTIVES:

I. To evaluate, in previously untreated patients with high risk (IPI 3-5) DLBCL treated with rituximab intense dosing and CHOP-21: Complete response (CR) rate, (as defined by International Harmonization Project criteria using 18-fluorodeoxyglucose [FDG] -positron emission tomography [PET]/computed tomography [CT]).

II. Overall survival.

III. Toxicity profile.

IV. Rituximab pharmacokinetics for this dose and schedule.

V. Effect of immunophenotype of DLBCL on outcome.

VI. Effect of Fc-Gamma Receptor III (FcyRIII) polymorphism genotype on outcome. OUTLINE: Patients receive rituximab intravenously (IV) on days 0, 1, 4, 8, and 15 of course 1; days 1, 8, and 15 of course 2; and day 1 of all subsequent courses. Patients also receive CHOP chemotherapy comprising cyclophosphamide IV, doxorubicin hydrochloride IV, and vincristine sulfate IV on day 1, and prednisone orally (PO) on days 1-5. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed up every 2-3 months for 2 years, every 6 months for 3 years, annually for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed cluster of differentiation (CD) 20+ DLBCL with IPI between 3-5
* No prior chemotherapy, radiation therapy or immunotherapy for DLBCL; a short course (< 2 weeks) of corticosteroids is allowed for symptom control Signed informed consent
* Eastern Cooperative Oncology Group (ECOG) Performance status assessed between 0 and 2; performance status of 3 will be accepted if impairment is caused by DLBCL complications and improvement is expected once therapy is initiated
* Measurable disease by Non-Hodgkin's Lymphoma Response Criteria on FDG-PET/CT; baseline measurements and evaluations must be obtained =< 21 days prior to registration
* Absolute neutrophil count (ANC) >= 1,500/μL unless due to marrow involvement by lymphoma
* Platelets >= 75,000/μL unless due to marrow involvement by lymphoma Hemoglobin > 7.0 g/dL unless due to marrow involvement by lymphoma
* Creatinine =< 2.0 mg/dL or calculated creatinine clearance >= 40
* Total bilirubin =< 1.5 mg/dL unless due to Gilbert's disease
* Aspartate aminotransferase (AST)/ alanine aminotransferase (ALT) =< 2.5 the upper limit of normal
* Alkaline phosphatase =< 5x upper limit of normal
* Patients with bilirubin between 1.5-3.0 mg/dL due to lymphoma may be entered and doses adjusted
* Left ventricular ejection fraction (LVEF) >= 50%

Exclusion Criteria:

* Women who are pregnant or breast feeding
* Known seropositivity for human immunodeficiency virus (HIV)
* Known presence of central nervous system (CNS) involvement by lymphoma
* New York Heart Association Classification III or IV heart
* Current or chronic hepatitis B or hepatitis C infection (as detected by positive testing for Hepatitis B surface Antigen [Hbs Ag] or antibody to Hepatitis C virus [anti HCV] respectively); patients must be tested for Hepatitis B surface antigen and anti-HCV =< 21 days prior to registration
* Male patients (with female sexual partners of childbearing potential) and female patients of childbearing potential who refuse to use effective methods of contraception
* Unstable or severe uncontrolled medical, psychological, or social condition
* Any evidence of serious active, uncontrolled infection (i.e., requiring an IV antibiotic or antiviral agent)
* Receipt of live vaccine within 4 weeks prior to study drug administration
* Concurrent active malignancy other than non-melanoma skin cancer or carcinoma in situ of the cervix; subjects with previous malignancies are eligible provided that they have been treated with curative intent and remain disease free for 3 years or more
* No prior chemotherapy for lymphoma
* Prior radiation therapy for lymphoma
* Any important medical illness or abnormal laboratory finding that would, in the investigator's judgment, significantly increase the subject's risk of participating in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
PFS following treatment with rituximab intense dosing and CHOP-21 in previously untreated patients with high risk DLBCL | 1 year
  Defined as the time from entry onto study until lymphoma progression or death from any cause.

SECONDARY OUTCOMES:
CR in previously untreated patients with high risk DLBCL treated with rituximab intense dosing and CHOP-21 | Baseline, between days 15 and 21 of course 3, and within 20-35 days after completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael Millenson, MD, FACP, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States